CLINICAL TRIAL: NCT05745909
Title: Randomized Single Center Clinical Trial Comparing Loop Ileostomy Versus Loop Transverse Colostomy in Patients After Major Anterior Resections
Brief Title: Trial Comparing Loop Ileostomy Versus Loop Transverse Colostomy
Acronym: LIVELOC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Republican Clinical Oncological Dispensary, Ministry of Health of the Republic of Bashkortostan (Other)
Responsible Party: Principal Investigator, Maksim Popov, Principal Investigator, Republican Clinical Oncological Dispensary, Ministry of Health of the Republic of Bashkortostan
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IK-001
Record Dates: First submitted 2023-02-04; First posted 2023-02-27 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Rectal Neoplasms; Ostomy; Neoplasms
Keywords: Rectal cancer; Low anterior resection; Loop transverse colostomy; Loop ileostomy; Stoma site infections
MeSH Terms: conditions — Rectal Neoplasms; Neoplasms | interventions — Laparoscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Loop transverse colostomy (Active Comparator): Laparoscopic or open low-anterior resection of the rectum with total mesorectal excision and created loop transverse colostomy
  Interventions: Procedure: Laparoscopic or open low-anterior resection of the rectum with TME and created loop transverse colostomy
- Loop ileostomy (Experimental): Laparoscopic or open low-anterior resection of the rectum with total mesorectal excision and created loop ileostomy
  Interventions: Procedure: Laparoscopic or open low-anterior resection of the rectum with TME and created loop ileostomy

INTERVENTIONS:
Procedure: Laparoscopic or open low-anterior resection of the rectum with TME and created loop transverse colostomy — The loop transverse colostomy is matured without torsion using a plastic retainer. The stoma protrudes 2-3 cm. The loop of the transverse colon is sutured with interrupted sutures using an absorbable 3/0 polyglactin suture without piercing the intestinal wall. The intestinal lumen is opened through a transverse incision on the antimesenteric border.
  Arms: Loop transverse colostomy
Procedure: Laparoscopic or open low-anterior resection of the rectum with TME and created loop ileostomy — The loop ileostomy is matured 25-30 cm from the ileocecal angle without torsion and without a retainer, so that stoma protrudes 2-3 cm. The loop of the ileum is sutured with interrupted sutures using an absorbable 3/0 polyglactin suture without piercing the intestinal wall. The intestinal lumen is opened through a transverse incision on the antimesenteric border.
  Arms: Loop ileostomy

SUMMARY:
The purpose of this study is to determine which stoma creation technique is preferable after low anterior resection of the rectum.

DETAILED DESCRIPTION:
The investigators enroll patients with a histologically confirmed diagnosis of primary rectal cancer with or without prior chemoradiotherapy who were hospitalized at the Ufa Republican Clinical Oncology Center from February 2023 to February 2024.

All patients undergo planned laparoscopic or open low-anterior resection of the rectum with total mesorectal excision. Patients are randomized into 2 groups in a 1:1 ratio. In the first group, a loop transverse colostomy is created, and in the second group, a loop ileostomy is created. The stoma exit sites are marked in advance the day before the surgery. The bowels are prepared by mechanical means (a polyethylene glycol-based laxative with a cleansing enema) according to a standard procedure before the surgery. Standardized stoma creation techniques are used. The resected parts are collected through a separate access. Patients are followed up for 60 days after surgery.

The sample size should be 124 patients to reach statistical significance (α = 0.05, study power 80%, confidence interval (CI) = 95%.). Considering possible losses during the study, the number of patients was increased to 130.

The investigators hypothesis is that the loop ileostomy group has a 20% higher incidence of stoma dysfunction but a 20% lower incidence of SSI (stoma site infections) compared to the loop colostomy group.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed adenocarcinoma of the rectum (stages 1-3 according to MRI)
* ECOG status 0-2,
* ASA≤3.
* At least 18 years of age
* Written informed consent

Exclusion Criteria:

* Emergency surgery;
* Previously formed stoma;
* Stage 4 disease;
* Obstructive resection of the rectum;
* Patients older than 79 years

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2023-03-01 (Actual); Primary Completion 2024-05-31 (Actual); Study Completion 2024-07-30 (Actual)

PRIMARY OUTCOMES:
SSI | 60 days after surgery
  incidence of stoma site infections
Ileus | 60 days after surgery
  incidence of stoma dysfunction

SECONDARY OUTCOMES:
Readmission rate | within the first 60 days after surgery
  readmission rate
Length of hospital stay | From date of surgery until the date of discharge, assessed up to 60 days
  the number of days from surgery to discharge
Time to stoma closure | within the first 6 months days after surgery
  the number of days from surgery to stoma closure
Time to first stool | 60 days after surgery
  the occurrence of anything other than serous-hemorrhagic contents in the colostomy bag
Time to adjuvant postoperative chemotherapy | within the first 2 months days after surgery
  the number of days from surgery to hospitalization for first chemotherapy
Quality of life in patients with ostomy | within the first 60 days after surgery
  estimated using EORTC QLQ-CR29

CONTACTS AND LOCATIONS:
Locations (1):
- Republican clinical oncological dispencery, Ufa, Bashkortostan Republic, Russia